CLINICAL TRIAL: NCT06269874
Title: A Single-centric, ProspectivE, Randomized Controlled Study Comparing Two Administration Pathways for Adenosine During Invasive Assessment of Microvascular Function in Patients With ANOCA.
Brief Title: Study Comparing Two Administration Pathways for Adenosine During Microvascular Function Assessment
Acronym: ASPERA-ANOCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tommaso Gori, Professor, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ASPERA-ANOCA; 20240124 (Other: JohannesGU)
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Microvascular Coronary Artery Disease
Keywords: adenosine; coronary microvascular assessment; microvascular disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to one of the two study arms and then the following study procedures will repeated in cross-over. Randomization will be done by using a computer-generated random sequence (medcalc, mariakerke, BE).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcome assessors will be blinded to the randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Adenosine (Active Comparator): Invasive microvascular function assessment will be conducted by administering intravenous hyperemic agent adenosine.
  Interventions: Diagnostic Test: microvascular function assessment
- Intracoronary Adenosine (Experimental): Invasive microvascular function assessment will be conducted by administering intracoronary hyperemic agent adenosine.
  Interventions: Diagnostic Test: microvascular function assessment

INTERVENTIONS:
Diagnostic Test: microvascular function assessment — mircovascular function parameters will be measured by administering adenosine in two different pathways

SUMMARY:
The aim of this study is to investigate the agreement and reproducibility between intravenous and intracoronary adenosine administration during invasive assessment of microvascular function.

Goals of this study are:

1. Agreement and reproducibility between intravenous and intracoronary adenosine administration in the IMR (Index of microvascular resistance) value.
2. Agreement and reproducibility of FFR(fractional flow reserve), CFR (coronary flow reserve), MRR (microvascular resistance reserve), RRR (resistive reserve ratio) and reproducibility of each of these as compared with CFRabs (absolute coronary flow).
3. Time required for IMR measurements

DETAILED DESCRIPTION:
The study is a single-center randomized, cross-over controlled, open label trial to investigate the reproducibility and agreement between intravenous and intracoronary adenosine administration during invasive assessment of microvascular function.

The primary analysis will be on the per-protocol population (i.e. including all patients who are not protocol violators).

Primary endpoint:

1. Agreement and reproducibility between intravenous and intracoronary adenosine administration in the IMR value.

Secondary endpoints:

1. Agreement and reproducibility of FFR, CFR, MRR, RRR and reproducibility of each of these as compared with CFRabs.
2. Time required for IMR measurements
3. Presence and severity of angina, assessed by SAQ(Seattle Angina Questionnaire)-7
4. Assessment of safety: Presence and severity of AV( atrioventricular) block, dyspnea, flush

ELIGIBILITY:
Inclusion Criteria:

* Chronic coronary syndrome (including patients with anginal equivalents).
* Indication to cardiac catheterization;
* Indication to the assessment of microvascular function (note: patients will be asked for participation and consented prior to the first measurement of microvascular function, which will be conducted as per clinical indication)
* Willingness to participate and ability to understand, read and sign the informed consent
* Age>18 years

Exclusion Criteria:

* Age <18 years
* Bronchial asthma, COPD (chronic obstructive pulmonary disease)
* Secondary or tertiary atrioventricular block without prior pacemaker implantation
* Previous CABG (coronary artery bypass graft) with patent grafts to the left anterior descending coronary
* Epicardial coronary disease (FFR <0.80 with evidence of a focal stenosis) in the left anterior descending territory
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2027-03-02 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between intravenous and intracoronary adenosine responses (IMR) | 6 months
  Agreement and reproducibility between IMR (index of microvascular resistance) obtained with intravenous and intracoronary adenosine administration during invasive assessment of microvascular function as assessed by Cohen´s Kappa, intraclass correlation coefficient and Bland-Altman analysis.

SECONDARY OUTCOMES:
Agreement between secondary parameters and reproducibility as compared with absolute | 6 months
  Agreement and reproducibility between secondary parameters (MRR, RRR, Pd/Pa, FFR, CFR, Ach-IMR) obtained with intravenous and intracoronary adenosine administration during invasive assessment of microvascular function as assessed by Cohen´s Kappa, intraclass correlation coefficient and Bland-Altman analysis.
Time required for IMR measurements | 6 months
  Comparison of time required for measuring IMR between intracoronary and intravenous adenosine administration

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Gori, MD,PhD, Principal Investigator — Center of Cardiology, Cardiology I, University Medical Center Mainz
Locations (1):
- Center of Cardiology, Cardiology I, university hospital Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No